CLINICAL TRIAL: NCT01035476
Title: Effectiveness Trial of Detailed NIPPV Feedback to Patients
Brief Title: Optimizing NIPPV Use for Patients With ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ALSA-P-2008-09
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: ALS
Keywords: ALS; nasal ventilation; data card recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Data Card Report (Experimental): Patients receive detailed reports of acceptance and adherence, with linked recommendations to optimize NIPPV.
  Interventions: Behavioral: Data Card Report
- Standard NIPPV Care (No Intervention): Patients receive routine monitoring and care related to NIPPV.

INTERVENTIONS:
Behavioral: Data Card Report — Patients received detailed report of acceptance and adherence base don data card information, with linked recommendations, to optimize use.
  Arms: Data Card Report

SUMMARY:
This research will examine the utility of the data card recording capacity of nasal ventilation devices (NIPPV) in people with ALS to optimize use.

DETAILED DESCRIPTION:
The data card records critical features of NIPPV acceptance (hours and timing of use) and adherence (apnea/hypopnea index, mask leak, minute ventilation); but to date data card monitoring has not yet been incorporated fully into ALS clinic practice. We will limit our focus to patients who meet Medicare-reimbursement criteria or AAN-recommended practice parameters for initiating NIPPV. The larger question guiding this research is whether data card monitoring and communication of these results to clinicians and patient families promotes "optimal use" of NIPPV. We define optimal use as (i) high acceptance, as indicated by daily night time use greater than 4 hours, and (ii) high adherence, as indicated by apnea/hypopnea index, mask leak, and minute ventilation. We will test whether timely reporting of acceptance and adherence values to patients and clinicians increases the likelihood of (i) changes in orofacial masks and settings on devices and continued use of devices, and (ii) positive patient mood and sleep quality and lower caregiver burden over follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable ALS
* Medicare or AAN criteria for initiating NIPPV
* Community resident
* English speaker

Exclusion Criteria:

* Unable to give informed consent
* Other pulmonary or cardiac conditions that complicate use of NIPPV
* Report from physician that participation would be harmful

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Length of time on NIPPV | 6 months

SECONDARY OUTCOMES:
Patient sleep quality, mood, fatigue | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Albert, PhD, Principal Investigator — University of Pittsburgh; David Lacomis, MD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States